CLINICAL TRIAL: NCT07142694
Title: Evaluation of a Plant-based Protein Pudding In Older Adults Attending a Medically Managed Fitness Facility
Brief Title: Feasibility of Adding a Plant-Based Protein Pudding to the Diet of Older Adults Who Attend a Medically Managed Fitness Facility
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seven Oaks Hospital Chronic Disease Innovation Centre (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HS26887 (B2025:025)
Record Dates: First submitted 2025-07-10; First posted 2025-08-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Feasibility Studies; Nutrition Intervention

STUDY DESIGN:
Intervention Model Description: This trial is a randomized controlled parallel arm feasibility trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant Based Pudding (Experimental): Participants will consume plant based pudding daily for 7 days per week
  Interventions: Dietary Supplement: Plant Based pudding
- Continue with their current lifestyle (No Intervention): Participants will continue with their current lifestyle without intervention

INTERVENTIONS:
Dietary Supplement: Plant Based pudding — Will consume one high protein plant based pudding daily for 7-days per week for 12 weeks
  Arms: Plant Based Pudding

SUMMARY:
The goal of this a 12-week randomized controlled parallel arm feasibility trial is to evaluate the feasibility and acceptability of incorporating a plant-based protein pudding into the diets of older adults who attend a medically managed fitness facility. The primary participant population includes older adults, aged 60 years and above, who are generally healthy and engaged in structured fitness programs.

The main questions it aims to answer are:

Is a plant-based protein pudding acceptable and well-tolerated by older adults? Does regular consumption of the pudding support muscle health and overall well-being in this population?

Participants will:

Consume a plant-based protein pudding as one arm daily for 7 days per week (experimental) and the other will continue their current lifestyle (control).

The experimental group will complete surveys or questionnaires to assess acceptability, taste, and ease of integration into daily meals.

Undergo basic physical or health assessments (e.g., muscle function or strength evaluations) to evaluate potential effects.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial
* Male or female aged ≥60 years
* Actively attend the Wellness Institute (≥8 times in the past 28 days),

Exclusion Criteria:

* Allergy to ingredients in the study treatment
* Inability to consume treatment product
* Inability to obtain written informed consent
* Apart of any physical rehab program at WI (cardiac rehab, kidney fit, etc. )

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Eligibility to Randomization Ratio for Feasibility | Measured upon study completion after 12-weeks
  A ratio of eligibility to randomization will be collected at 12 months. The trial will be considered feasible if ratio falls within >0.5, calculated as the ratio of individuals who were randomized to the trial to the number eligible to participate who were approached to participate.
Recruitment Rate | during 12 months
  Recruitment rate will be assessed as the average number of new participants enrolled per site per week during the active recruitment period, with a target of ≥0.5 participants per site per week.
Follow up rate | Measured at end of 12 weeks
  Follow-up rate (% of participant outcomes) will be calculated if more than >85% of participant outcomes
Adherence to Intervention | Measured at the end of 12 weeks
  Adherence to plant based pudding intervention if more than (75% of dispensed plant based pudding protein is consumed)

SECONDARY OUTCOMES:
Serum Pre-Albumin | Measured at Baseline Week 1 and at the end of 12 weeks.
  Serum albumin is measured in grams per deciliter (g/dL)
Blood Amino Acid Profile | Measured at Baseline Week 1 and at the end of week 12
  blood amino acid profile
Dry Weight | Measured at Baseline Week 1 and after the end of week 12
  Changes in body weight (Kg)
Waist Circumsference | Measured at Baseline Week 1 and after the end of week 12
  Measured in cm
Lean mass | At the baseline week 1 and at end of week 12
  Measured in Kg
Fat Mass | At the baseline week 1 and at end of week 12
  Measured in Kg
Physical function; Five rep chair stand time test | Measured at Baseline Week 1 and after the end of week 12
  the amount of time it takes for a participant to get up out of a chair five times measured in seconds
Blood Pressure | Measured at Baseline Week 1 and after the end of week 12
  Systolic and Diastolic Blood Pressure Measured in mmHg
Total Calories intake | Measured at Baseline Week 1 and after the end of week 12
  Using RxFoods- Diet recall change in total calories measured in kcal/day
Carbohydrates | At the baseline week 1 and at end of week 12
  Measured as g/day
Protein | At the baseline week 1 and at end of week 12
  Measured as g/day
Fat | At the baseline week 1 and at end of week 12
  Measured as g/day
Fiber (total dietary fiber) | At the baseline week 1 and at end of week 12
  Measured as g/day

CONTACTS AND LOCATIONS:
Locations (1):
- Chronic Disease Innovation Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No